CLINICAL TRIAL: NCT06385015
Title: Targeted Upstream Prevention (T-UP): Engaging Vulnerable Students in Diabetes Prevention
Brief Title: T-UP: Engaging Vulnerable Students in Diabetes Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Lauren Wisk, PhD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB#23-001257
Record Dates: First submitted 2024-01-23; First posted 2024-04-25 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2; PreDiabetes
Keywords: Prediabetes; Type 2 Diabetes; Diabetes Prevention Program
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Prevention Program (DPP) group (Experimental): The DPP group will receive a tailored Diabetes Prevention Program.
  Interventions: Behavioral: Tailored DPP Intervention
- Control group (No Intervention): The control group will receive access to materials on study habits (fall), alcohol use (winter), and financial literacy (spring). The control group will receive the materials via e-mail for participants to review on their own time. A research assistant will meet with control participants via Zoom to explain the materials. The Zoom session will take approximately 1 hour.

INTERVENTIONS:
Behavioral: Tailored DPP Intervention — The intervention includes 19 sessions (18 in-person and 1 on-demand) covering 24 DPP modules; each session is approximately an hour in length and will be moderated by a trained lifestyle coach. Lifestyle coaches are accessible, collaborative, and culturally competent diabetes care and education specialists trained and certified in the CDC's National DPP curriculum to provide effective guidance and support for program participants. Each group will meet regularly during the academic year, with six in-person sessions delivered per 10-week quarter (for each of three quarters) to allow for breaks during final exams and scheduled school recess (e.g., spring break). It will take place on UCLA campus.
  Arms: Diabetes Prevention Program (DPP) group

SUMMARY:
The goal of this study is to enhance reach and uptake of diabetes prevention among young adults, with a focus on recruiting underserved and high-need students who face additional challenges, including food and financial insecurity.

The specific aims are to: 1) Evaluate the efficacy of adolescents and young adults (AYA)-tailored version of the University of California Diabetes Prevention Program (UC DPP) for mitigating type 2 diabetes risk (i.e., weight change) in a pre/post pilot trial. The investigators hypothesize that the AYA-tailored intervention will be effective at producing 5% weight loss from baseline to program completion (at 9-months); and, 2) Assess the feasibility and acceptability of an AYA-tailored version of the UC DPP program. The investigators hypothesize that it will be feasible to recruit the desired number of participants given proposed innovative outreach strategies, and that the AYA-tailored intervention will be deemed acceptable to participants both qualitatively and in regards to their retention in the program at rates similar to the larger UC DPP.

The investigators will randomize participants to the AYA-tailored DPP cohort vs control cohort. Control participants will be offered the opportunity to participate in the AYA-tailored DPP in the following academic year. Participants will be organized into groups within their DPP cohort based on their student status and/or place of residence. The intervention will include 19 sessions (18 in-person and 1 on-demand) covering 24 DPP modules; each session is approximately an hour in length and will be moderated by a lifestyle coach. At the end of each session, intervention participants will receive an email/text with a unique link to a brief REDCap survey to ascertain acceptability of the session. Control group will receive access to materials about study habits, alcohol use, and financial literacy. Control group will receive materials via e-mail for participants to review on their own time and will receive acceptability surveys. A research assistant (RA) will meet with control participants via Zoom to explain the materials. Participants will complete baseline and 9-month follow-up assessments. Participants will complete a 30 minute questionnaire via REDCap and height/weight measurements will be collected by a RA. Participants will be asked to self-report weight and physical activity at the end of the fall and winter quarter; data will be collected via brief REDCap survey.

DETAILED DESCRIPTION:
Aim 1 - Design: Pre/post pilot trial of 100 participants (<1% of total number of eligible UCLA undergraduates). The investigators will randomize participants to the AYA-tailored DPP vs control based on a stratified, block (n=2) schema based on age [≤19/≥20] and sex [M/F]. All control participants will be offered the opportunity to participate in the AYA-tailored DPP in the following academic year (in the interest of equipoise).

Aim 1 - Participant Recruitment: All participants will be asked to complete a brief online intake form to assess eligibility and to collect preferred contact information. This form will further allow the investigators to prioritize recruitment efforts of those with identified food, financial, or stress-related vulnerability (per standard NCHA questions). After confirming eligibility, a trained research assistant (RA) will reach out to eligible participants to obtain informed consent and enroll them in the pilot trial.

Aim 1 - Tailored DPP Intervention: Once consented and enrolled, participants will be randomized into one of two cohorts, the first group will be enrolled in the tailored DPP for the immediate academic year while the second will be enrolled in a series of unrelated interventions in year 1 and offered the opportunity to participate in the AYA-tailored DPP for the following academic year. As social support is a key component of the program, participants will be organized into groups within their DPP cohort based on their student status (frosh/soph vs junior/senior) and/or place of residence (residence hall vs off-campus). The intervention will include 19 sessions (18 in-person and 1 on-demand) covering 24 DPP modules; each session is approximately an hour in length and will be moderated by a trained lifestyle coach. Lifestyle coaches are accessible, collaborative, and culturally competent diabetes care and education specialists trained and certified in the CDC's National DPP curriculum to provide effective guidance and support for program participants. The Lifestyle Coach's ability to support participants, provide guidance, and help groups work together effectively is essential for a successful lifestyle change program. Each group will meet regularly during the academic year, with six in-person sessions delivered per 10-week quarter (for each of three quarters) to allow for breaks during final exams and scheduled school recess(e.g., spring break). The interventions for the intervention participants will take place on UCLA campus. It will take place at the John Wooden Center, UCLA Teaching Kitchen, UCLA dining halls, UCLA sculpture garden, UCLA botanical garden, UCLA Arthur Ashe Student Health & Wellness Center, UCLA Glendon building, UCLA Murphy Hall, and other UCLA buildings. UC DPP has consistently been using some of these places to facilitate the program.

The control group will receive access to a study habits intervention (fall), alcohol use intervention (winter), and financial literacy intervention (spring). The control group will receive each intervention materials via e-mail for participants to review on their own time. The interventions for the control group will be remote. A research assistant will meet with control participants via Zoom to explain the intervention materials. The Zoom session will take approximately 1 hour. At the end of each session, participants will receive an email or text (depending on their preferred method of contact) with a unique link to a brief (~1 minute) REDCap survey to ascertain acceptability of the session. There will be three zoom sessions in total (one for each intervention).

The last acceptability survey of the Fall and Winter quarter for the intervention group (and the only acceptability survey for the control group) will ask about self-reported weight and physical activity. The investigators will send the last acceptability survey of the Fall and Winter quarter for the intervention group around the same time the investigators will send the only acceptability survey for the control group.

Aim 1 - Data Collection: Participants will complete two study assessments (baseline and 9-month follow-up).There are two assessments per year, baseline and 9-month follow up for the first year and baseline and 9-month follow-up for the second year. These assessments will be done in October and June, respectively. Participants will complete a 30 minute questionnaire (administered as a Research Electronic Data Capture (REDCap) survey) and height/weight measurements will be collected using a standardized protocol by a trained research assistant. RA will meet participants at the Wooden Center to collect measurements. Participants will be asked to self-report weight and physical activity at the end of the fall and winter quarter; data will be collected via brief REDCap survey.

Aim 1 - Measures: The baseline survey assessment will collect data using validated tools on sociodemographics (e.g., age, sex, race, ethnicity, socioeconomic status), social vulnerability (food security using the USDA ERS Food Security 6-Item Short Form, financial security using the Financial Chronic Stress Scale), health-related quality of life (CDC's HRQoL tool), mental health (depressive symptoms via Patient Health Questionnaire-8; anxiety symptoms via Generalized Anxiety Disorder-7), self-perceived weight status (How do you describe your weight?), and self-reported physical activity and diet (using the International Physical Activity Questionnaire and Nutrition Screening Survey). Follow-up assessment (at 9 months) will collect data on health-related quality of life, mental health, self-perceived weight status, and self-reported physical activity and diet. At both time points, height and weight data will be collected by a trained research assistant.

Aim 2 - Design: Longitudinal analysis of participants of the treatment arm (N=50 in the AYA-tailored DPP cohort).

Aim 2 - Data Collection: At the end of each session, participants will receive an email or text (depending on their preferred method of contact) with a unique link to a brief (~1 minute) REDCap survey to ascertain acceptability of the session. Intervention participants will be asked to complete at least 15 out of the 18 acceptability surveys. The investigators will implement targeted follow-up reminder schemes via text-messaging and/or e-mail, to improve participant response rates to these brief interim assessments.

Aim 2 - Measures: To assess feasibility the investigators will determine proportion of participants who are recruited (enrolled /those completing the initial screen) and retained (session completion / enrolled). Recruitment source (student health referral vs diffuse outreach/self-referral) will be compared to determine if characteristics of participants differed by recruitment source. Acceptability surveys will ask participants to rate satisfaction with each session on a 5-point Likert scale ("very dissatisfied" to "very satisfied") with respect to a) content, b) coach, c) group interaction, and d) overall. Surveys will include an open-ended question to elicit participants' specific thoughts/perspectives on each session. Retention will be ascertained via attendance taken by the lifestyle coach.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are currently enrolled (either full time or part time) as an undergraduate at UCLA and meet criteria for the T-UP Wellness Program (students who have a BMI of ≥25 (≥23 for those self-identifying as Asian) and either documented prediabetes or identified as high-risk on a CDC questionnaire)

Exclusion Criteria:

* Participants who are not currently enrolled (either full time or part time) as an undergraduate at UCLA and do not meet criteria for the T-UP Wellness Program.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Change in weight (pounds, lbs) between baseline and 9-month follow-up | 9 months
  A physical scale will be used to assess the percent weight (in pounds) at baseline and at 9-months follow-up; change in these two measures will be calculated and used as the primary outcome. The investigators are comparing the percentage change between participants' final weight (in pounds) measurement versus baseline weight (in pounds) measurement as a fraction of participants' baseline weight measurement (= (final - baseline) / baseline)).
Change in self-reported quality of life (Centers for Disease Control and Prevention Health-Related Quality of Life-14 item (CDC HRQOL-14)) between baseline and 9-month follow-up | 9 months
  A self-reported questionnaire will be administered at baseline and 9-month follow-up and will include questions from the three different modules of the CDC HRQOL-14. The summary "unhealthy days" index, which ranges from 0-30 unhealthy days, will be calculated. Higher scores indicate worse health/well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Wisk, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will add data resources to figshare (https://figshare.com/), an ADA and NIH approved general data repository. The data repository will include the data codebook and information to submit a reasonable request for data access. Reasonable request will be one that meets the following criteria: submitted by a credentialed (professional/graduate degree holder or student) researcher affiliated at a college, university, medical center/system or other non-profit institution, with a proposed research question that is addressable with the available data (regardless of the perceived merit of the question), who is willing to agree to cite the original data source and ADA as a funding source for all research products using the data, and who is willing to agree to not attempt to identify any of the participants included in the dataset. Once a reasonable request has been submitted, the investigators will provide aggregate, de-identified study data to researchers.
Time Frame: The data dictionary/codebook and request instructions will be made available 6 months after the completion of data collection and cleaning.
Access Criteria: A credentialed researcher affiliated at a college, university, medical center/system or other non-profit institution, with a proposed research question that is addressable with the available data, who is willing to agree to cite the original data source and ADA as a funding source for all research products using the data, and who is willing to agree to not attempt to identify any of the participants included in the dataset.

DOCUMENTS (1):
  • Informed Consent Form (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT06385015/ICF_000.pdf